CLINICAL TRIAL: NCT00158054
Title: Consortium for Translation of Psychosocial Depression Theories to Interventions and Dissemination - Project 2: Phase I Randomized Controlled Trial of Patient Preference, Stepped-Care Treatment For Distress in Heart Disease Patients
Brief Title: COPES Phase I Randomized Controlled Trial of Treatment For Distress in Heart Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Karina Davidson, Professor of Behavioral Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAB5166; GCO 02-0247 (Other: Grant ID); N01HC25197-0-0-0 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Heart Diseases; Depression
Keywords: depression; acute coronary syndrome; clinical trials
MeSH Terms: conditions — Heart Diseases; Depression; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Condition (INT) (Experimental): Enhanced depression care: Participants assigned to INT condition will be given an information brochure describing the intervention. This description will include an overview of the two elements of treatment (Problem Solving Therapy (PST), pharmacotherapy), the choice that the participant has for which element of treatment they will receive, and the stepped care aspect of treatment.
  Interventions: Behavioral: Enhanced depression care
- Usual Cardiologic Care Condition (UCC) (Other): Referred depression care: Participants assigned to the usual cardiologic care condition (UCC) condition will be scheduled for their next follow-up visit and thanked for their time.
  Interventions: Behavioral: Referred depression care

INTERVENTIONS:
Behavioral: Enhanced depression care — Initial patient preference for problem-solving therapy and/or pharmacotherapy, then a stepped-care approach.
  Other Names: Patience-preference; stepped care distress treatment; intervention condition (INT)
  Arms: Intervention Condition (INT)
Behavioral: Referred depression care — Physician notified of depression symptoms, usual care followed.
  Other Names: Usual Cardiologic Care (UCC)
  Arms: Usual Cardiologic Care Condition (UCC)

SUMMARY:
The specific aim of the "Coronary Patients Evaluation Study" (COPES) Project 2 is, within a Phase-I RCT, to examine patient satisfaction, treatment safety, and symptom reduction associated with treatment for symptoms of distress and/or depressed mood among post acute coronary syndrome (ACS) patients, as compared to usual cardiology care. For the purposes of this study, "symptoms of distress and/or depressed mood" is defined by a score on the Beck Depression Inventory (BDI) >10. The specific treatment approach utilized follows the, "Improving Mood-Promoting Access to Collaborative Treatment" (IMPACT) Clinical Trial, and involves up to 6-months of a patient preference, stepped-care protocol. Within this protocol, patients choose between brief, problem focused psychotherapy and anti-depressant medication. Treatment progress is reviewed at 2-month intervals, providing opportunities to 'step-up' treatment if patients are not demonstrating sufficient symptom reduction.

DETAILED DESCRIPTION:
Objectives: To examine patient satisfaction, treatment safety, and symptom reduction associated with treatment for symptoms of distress and/or depressed mood among post acute coronary syndrome (ACS) patients, as compared to usual cardiology care.

Research Design: The Study utilizes a Phase-I RCT design to achieve this Aim.

Methodology: Patients with confirmed ACS are screened for symptoms of distress and/or depressed mood within 7 days of the index ACS event, using the Beck Depression Inventory (BDI). Those meeting inclusion criterion on the BDI (score>10) and consenting to study are followed for 3-months, at which time they are re-assessed. Those continuing to show BDI score >10 and consenting, are randomized to the intervention condition (INT) or to usual cardiologic care (UCC). INT is defined by up to 6-months of a patient preference, stepped care treatment whereby patients chose between brief, problem-focused psychotherapy (PST) and antidepressant medication (MED). Patients are re-evaluated at 2- and 4-months after randomization. Those not showing sufficient improvement in symptoms receive augmented therapy. Those who initially choose PST can receive more frequent sessions and/or the addition of MED; those who initially choose MED can receive a change of agent, an increase in dosage, an additional medication, and/or PST.

Hypotheses to be tested are:

1. Patient satisfaction within intervention treatment (INT) will be higher than in the usual cardiologic care (UCC) condition, as evidenced by self-report and levels of participation
2. The INT group will experience a greater reduction in symptoms of distress and/or depression over the treatment period than the UCC group (secondary hypothesis).
3. Improvement in symptoms of distress and/or depression will be associated with reduction in levels of inflammatory markers and improvement in adherence with physician prescribed aspirin therapy (secondary hypothesis).

This is a multi-site study involving Mt. Sinai, and Yale and Columbia University Schools of Medicine. A total of 500 people will be screened into the initial 'observational period', which occurs at the time of new ACS diagnosis. From among these, it is anticipated that 200 people will evidence persistent BDI > 10 at 3-month follow-up and agree to be enrolled in the Phase 1 RCT.

The clinical relevance of the Study concerns demonstration of the acceptability and satisfaction with the treatment approach by post-ACS patients, as preliminary to a Phase-III RCT that would test the effect of such an intervention on event-free survival after ACS.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization with a verified diagnosis of unstable angina (UA) or acute myocardial infarction (AMI). UA is defined as new-onset angina within 2 months, exacerbation of previous angina with pain at rest or with minimal exercise, prolonged chest pain (lasting > 20 minutes), or angina within 2 weeks following discharge for myocardial infarction in patients with documented coronary artery disease (defined as ischemic ECG ST-T segment changes, previously documented MI, positive nuclear treadmill test result, or coronary angiographic evidence of blockage of 50% stenosis in >1 major coronary artery). AMI is defined as at least 2 of the following: ischemic chest pain lasting >20 minutes, acute rise in serum troponin-I >1.0 ng/L, and new pathologic ST segments in >2 contiguous ECG leads.
2. Score on the Beck Depression Inventory (BDI) > 10 within 7 days of index ACS event and 3-months later.

Exclusion Criteria:

1. active suicidal or homicidal ideation, as these patients require immediate referral for assessment and treatment (see below for procedures for these patients);
2. current alcohol or other substance abuse disorders (as depressive symptoms may be a result of these disorders),
3. any current psychotic disorder,
4. history of psychotic disorder, bipolar disorder, or serious personality disorders,
5. diagnosis of a terminal non-cardiac illness,
6. ACS diagnosis secondary to diagnosis of a severe medical disease,
7. inability to communicate in English,
8. levels of cognitive impairment indicative of dementia,
9. unavailability for the period of the study,
10. overt hypothyroid, and
11. currently taking triptans.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, Ph.D., Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Ye S, Shaffer JA, Rieckmann N, Schwartz JE, Kronish IM, Ladapo JA, Whang W, Burg MM, Davidson KW. Long-term outcomes of enhanced depression treatment in patients with acute coronary syndromes. Am J Med. 2014 Oct;127(10):1012-6. doi: 10.1016/j.amjmed.2014.05.004. Epub 2014 May 14. PMID 24835038
- [Derived] Davidson KW, Rieckmann N, Clemow L, Schwartz JE, Shimbo D, Medina V, Albanese G, Kronish I, Hegel M, Burg MM. Enhanced depression care for patients with acute coronary syndrome and persistent depressive symptoms: coronary psychosocial evaluation studies randomized controlled trial. Arch Intern Med. 2010 Apr 12;170(7):600-8. doi: 10.1001/archinternmed.2010.29. PMID 20386003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 hospital sites (Mount Sinai Hospital and New York Presbyterian Hospital, New York, New York; and New Haven Hospital, Hospital of St Raphael, and Veterans Affairs Connecticut Healthcare System-West Haven, New Haven, Connecticut) from January 1, 2005, through February 29, 2008.
Groups:
- Enhanced Depression Care: The intervention included the following 5 essential components adapted from the IMPACT study: (1) an enhanced care approach, with treatment delivered by a clinical nurse specialist, psychologist, social worker, and/or psychiatrist; (2) patient choice of psychotherapy and/or pharmacotherapy; (3) a form of psychotherapy called problem-solving therapy (PST); (4) a stepped-care approach in which symptom severity was reviewed every 8 weeks and treatment was augmented according to predetermined decision rules; and (5) a standardized instrument used to track depressive symptoms.
- Referred Depression Care: The control condition for the trial was usual care, as defined by the patient's treating physicians. Physicians of the usual care patients were informed that their patients were participating in a trial and that they had elevated depressive symptoms; physicians were also told whether the patient met the criteria for a major depressive episode.
Period: Overall Study
Arm/Group | Enhanced Depression Care | Referred Depression Care
Started | 80 | 77
Completed | 70 | 74
Not Completed | 10 | 3
Not completed — Refused to continue | 3 | 0
Not completed — Unavailable for follow up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Depression Care | Referred Depression Care | Total
Number analyzed (Participants) | 80 | 77 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.6) | 61.1 (10.6) | 60.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 39 | 34 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 32 | 68
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 47 | 40 | 87
  Black/African American | 12 | 17 | 29
  Asian/Indian | 8 | 7 | 15
  Asian/Pacific Islander | 0 | 1 | 1
  Native American | 1 | 0 | 1
  Other | 10 | 10 | 20
  Unknown/Decline to state | 2 | 2 | 4
Type of presenting acute coronary syndrome [Number; unit: participants] — MI = Myocardial Infarction
  participants
    Unstable angina | 58 | 60 | 118
    Non-ST-segment elevation MI | 13 | 9 | 22
    ST-segment elevation MI | 8 | 8 | 16
    Other | 1 | 0 | 1
Beck Depression Inventory Score, categorical [Number; unit: participants] — The Beck Depression Inventory (BDI) is a 21-item multiple choice, self-report instrument that is used to assess the severity of symptoms of depression. The score ranges from 0 (no symptoms) to 63 (worst symptoms).
  participants
    BDI score >=16 | 52 | 52 | 104
    BDI score < 16 | 28 | 25 | 53
Diagnosis of major depressive episode [Number; unit: participants]
  Yes | 23 | 21 | 44
  No | 57 | 56 | 113
GRACE ACS Risk and Mortality Score [Mean (Standard Deviation); unit: units on a scale] — The GRACE Risk and Mortality score is one tool used to help clinicians assess the future risk of death or myocardial infarction (MI), as a guide to treatment options, in a patient with an acute coronary syndrome (ACS).
  Range of values: 2 to 372. Patients are categorized as low risk (score <= 108), medium risk (score between 109 - 140), and high risk (>140 score).
  units on a scale | 91 (24) | 94 (23) | 93 (23)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Self-reported as Satisfied With Care for Depressive Symptoms.
Description: Number of participants who rated their depression care as excellent or very good as a percentage.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Enhanced Depression Care | Referred Depression Care
Number analyzed (Participants) | 80 | 77
percentage of participants | 54.2 | 18.8

2. Secondary Outcome: Level of Depressive Symptoms
Description: Depressive symptoms were measured using the Beck Depression Inventory (BDI), which is a 21-item multiple choice, self-report instrument that is used to assess the severity of symptoms of depression. The score ranges from 0 (no symptoms) to 63 (worst symptoms).
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Depression Care | Referred Depression Care
Number analyzed (Participants) | 80 | 70
units on a scale | 13.2 [11.1 to 15.3] | 17.7 [15.6 to 19.7]

3. Secondary Outcome: Number of Participants Experiencing Major Adverse Cardiovascular Events
Description: The table represents the number of participants experiencing major adverse cardiovascular events
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Enhanced Depression Care | Referred Depression Care
Number analyzed (Participants) | 80 | 77
participants | 3 | 10

4. Secondary Outcome: All-cause Mortality
Description: All- cause mortality
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Enhanced Depression Care | Referred Depression Care
Number analyzed (Participants) | 80 | 77
participants | 9 | 7

ADVERSE EVENTS:
Arm/Group | Enhanced Depression Care | Referred Depression Care
Serious Adverse Events (participants affected / at risk) | 22/80 | 22/77
Other Adverse Events (participants affected / at risk) | 60/80 | 74/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Depression Care (N=80) | Referred Depression Care (N=77)
ACS (intervention) (Cardiac disorders) | 5 | 7 — Acute coronary syndrome (intervention)
ACS (non-intervention) (Cardiac disorders) | 2 | 1 — Acute coronary syndrome (non-intervention)
Cath (diagnostic/non-intervention) (Cardiac disorders) | 1 | 4 — Catheterization (diagnostic/non-intervention)
Chest pain (Cardiac disorders) | 7 | 6
Chest pain (non-cardiac) (General disorders) | 1 | 1
Hypertension (Cardiac disorders) | 1 | 0
Hypotension/Postural Hypotension (Cardiac disorders) | 0 | 1
Intervention (scheduled/non-urgent) (Cardiac disorders) | 2 | 6
Life-threatening arrythmia (Cardiac disorders) | 1 | 1
Non-CV (General disorders) | 2 | 0 — Non-Cardiovascular
Other (cardiac) (Cardiac disorders) | 2 | 1
Other (non-cardiac) (General disorders) | 5 | 9
Other (psych) (Psychiatric disorders) | 1 | 0
Self-report only; no additional info (General disorders) | 1 | 1
Shortness of breath, fatigue, CHF (General disorders) | 2 | 4
Stroke (Vascular disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 1
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Depression Care (N=80) | Referred Depression Care (N=77)
Chest pain (Cardiac disorders) | 14 | 21
Chest pain (non-cardiac) (General disorders) | 4 | 8
Hypotension/Postural Hypotension (Cardiac disorders) | 1 | 1
Intervention (scheduled/non-urgent) (Cardiac disorders) | 0 | 1
Non-CV (General disorders) | 1 | 7 — Non-Cardiovascular
Other (cardiac) (Cardiac disorders) | 1 | 1
Other (non-cardiac) (General disorders) | 58 | 71
Other (psych) (Psychiatric disorders) | 47 | 62
Self-report only; no additional info (General disorders) | 1 | 5
Shortness of breath, fatigue, CHF (General disorders) | 23 | 34
Suicidal Ideation (Psychiatric disorders) | 7 | 11
Worsening Depressioin (Psychiatric disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No